CLINICAL TRIAL: NCT01422993
Title: A Pilot Study of a Strength and Balance Training Program for Persons With Oxaliplatin Induced Peripheral Neuropathy
Brief Title: Pilot Study of Strength and Balance Training Program for Persons With Oxaliplatin Induced Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: ONS Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-16557
Record Dates: First submitted 2011-08-23; First posted 2011-08-25 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Neuropathy; Gastrointestinal Cancer
Keywords: Oxaliplatin Induced; Peripheral Neuropathy; Strength; Balance; Training Program; Colon; Rectal
MeSH Terms: conditions — Gastrointestinal Neoplasms; Peripheral Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Excercise and Questionnaire (Experimental): 12 week exercise program followed by questionnaire.
  Interventions: Other: 12 Week Exercise Program

INTERVENTIONS:
Other: 12 Week Exercise Program — Participants will be asked to take part in a one hour exercise program twice a week for 12 weeks. They will also be asked to answer questionnaires and participate in an evaluation of their strength, balance, and physical function every 4 weeks immediately following the exercise program. This evaluation will take an additional hour every 4 weeks.

SUMMARY:
The purpose of this study is to evaluate the effects on strength, balance, and neuropathic symptoms (numbness, tingling, pain, weakness) of a 12 week, bi-weekly, 60 minute, group exercise program designed to improve lower extremity strength and balance with persons with oxaliplatin induced peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Prior history of colon cancer
* Completed oxaliplatin based chemotherapy at least 6 months prior to enrollment
* Report numbness, tingling, or pain of the lower extremities ≥ 4 by chemotherapy induced peripheral neuropathy (CIPN) Visual Analog Rating
* Karnofsky performance status of at least 60%
* Able to read, write, and understand English

Exclusion Criteria:

* Patients will be excluded from the study if they live outside of a 30 mile radius of the University of South Florida, if they are currently undergoing chemotherapy or radiation therapy, or if they regularly (at least once a week) participate in strength or balance training exercises. The investigators will not exclude participants if they are participating in aerobic exercise, but we will collect that information so that the investigators may control for aerobic exercise in our data analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-07; Primary Completion 2016-04 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of Screened Patients Who Participate and Complete the Study | 10 Months
  To evaluate feasibility, the percentage of patients screened to percentage enrolled in the study and the percentage enrolled to percentage that completes the study will be calculated. Patients who do not complete the study will be contacted to determine why they were unable to complete the study and the reasons will be recorded. How many sessions were attended will also be recorded.

SECONDARY OUTCOMES:
Number of Participants Who Experience Side Effects | 10 Months
  To evaluate tolerability, at each session, data regarding any participant who was unable to complete the entire session will be recorded along with any side effects that participants report. Participants will also be asked to rate the level of exercise they perform at each session as either a) too easy b) just right c) too challenging.
Number of Participants With Measured Improvement | 10 Months
  Treatment-effect size will be evaluated by means of changes in muscle strength, balance, and neuropathy from the beginning to completion of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Tofthagen, Ph.D., ARNP, Principal Investigator — University of South Florida
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States